CLINICAL TRIAL: NCT03366740
Title: Efficacy of GB Mixed Full Strength Rice Suji, and Full Strength Rice Suji Alone Compared to 3/4th Strength Rice Suji in the Management of PD in Children Aged > 6 Months to 36 Months: an Open-labeled Randomized Controlled Clinical Trial
Brief Title: Green Banana (GB) Mixed Diet in the Management of Persistent Diarrhea (PD)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PR-17075
Record Dates: First submitted 2017-11-05; First posted 2017-12-08 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2020-10

CONDITIONS: Persistent Diarrhea
Keywords: Persistent diarrhea; > 6 to 36 months aged children; green banana; rice suji; milk suji; comminuted chicken

STUDY DESIGN:
Intervention Model Description: Study design: This will be an open-labeled randomized controlled clinical trial with three treatment arms (3/4th strength rice suji, full strength rice suji with modification and GB mixed full strength rice suji). Investigators will prospectively screen, children > 6 to 36 months of age admitted to the Dhaka hospital of icddr,b, with PD or developed PD during their treatment period and failed to respond with milk suji and enroll them for the study. Thereafter permuted block randomization technique will be followed to select treatment arms for each child.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- GB mixed full strength rice suji (Experimental): On day 4 (3 days after milk suji) after diagnosis of PD, if PD doesn't resolve, the child will be enrolled in the study and after randomization will get the GB mixed full strength rice suji.
  The allocated diet will be continued for 7 days and a child will be followed. If there is deterioration of diarrhea (either increased frequency or watery consistency) for 3 days or condition remains static up to 7 days the child will be declared as treatment failure.
  Interventions: Other: GB mixed full strength rice suji
- Full strength rice suji alone (Experimental): On day 4 (3 days after milk suji) after diagnosis of PD, if PD doesn't resolve, the child will be enrolled in the study and after randomization will get full strength rice suji alone.
  Interventions: Other: Full strength rice suji Alone
- 3/4th strength rice suji (Active Comparator): On day 4 (3 days after milk suji) after diagnosis of PD, if PD doesn't resolve, the child will be enrolled in the study and after randomization will get 3/4th strength rice suji.
  Interventions: Other: 3/4th strength rice suji

INTERVENTIONS:
Other: GB mixed full strength rice suji — On day 4 (3 days after milk suji) after diagnosis of PD, if PD doesn't resolve, the child will be enrolled in the study and after randomization will get the Green banana mixed full strength rice suji The diet will be continued for 7 days and a child will be followed. If there is deterioration of diarrhea (either increased frequency or watery consistency) for 3 days or condition remains static up to 7 days the child will be declared as treatment failure.
  Arms: GB mixed full strength rice suji
Other: Full strength rice suji Alone — On day 4 (3 days after milk suji) after diagnosis of PD, if PD doesn't resolve, the child will be enrolled in the study and after randomization will get full strength rice suji alone.
  The diet will be continued for 7 days and a child will be followed. If there is deterioration of diarrhea (either increased frequency or watery consistency) for 3 days or condition remains static up to 7 days the child will be declared as treatment failure.
  Arms: Full strength rice suji alone
Other: 3/4th strength rice suji — On day 4 (3 days after milk suji) after diagnosis of PD, if PD doesn't resolve, the child will be enrolled in the study and after randomization will get 3/4th strength rice suji.
  The diet will be continued for 7 days and a child will be followed. If there is deterioration of diarrhea (either increased frequency or watery consistency) for 3 days or condition remains static up to 7 days the child will be declared as treatment failure.
  Arms: 3/4th strength rice suji

SUMMARY:
Diarrhea is the 2nd leading cause of death in under-five children. When diarrhea continued for 14 days or more it is known as Persistent Diarrhea (PD). In low and middle income countries (LMIC), 3%-23% of acute diarrheal episodes turn to PD. PD causes 32-62% of all diarrheal deaths in LMIC, and >25% in Bangladesh in contrast to 0.8% is caused by acute diarrhea. The prevalence of PD varied from 6.3 to 16.4 %. However, no larger prospective study was conducted to evaluate the efficacy of green banana in the management of PD among children older than 6 months.An open-labeled randomized controlled clinical trial is designed to assess the efficacy of green banana mixed full strength rice suji, and full strength rice suji alone compared to 3/4th strength rice suji in the management of persistent diarrhea (PD) in children aged > 6 months to 36 months in the Dhaka Hospital of icddr,b.

DETAILED DESCRIPTION:
Background:

Diarrhea, defined as passage of loose or watery stool 3 times or more in a 24 hour period, is the 2nd leading cause of death in under-five children. It accounts for 531,000 deaths among 5.9 million globally and 7,140 deaths among 119,000 Bangladeshi under-five deaths in 2015. Countries of Africa and South-East Asia, particularly India, Nigeria, Congo, Afghanistan, Pakistan, Ethiopia and Bangladesh face around 80% of total diarrhea related death of the world. Use of ORS and zinc reduced the number of diarrheal deaths, especially from acute diarrhea to 0.8%. However, when diarrhea continued for 14 days or more and which does not include recurrent or chronic diarrhea, such as coeliac disease, cystic fibrosis or congenital diarrheal disorders, it is known as persistent diarrhea (PD). In low and middle income countries 3%-23% of acute diarrheal episodes turn to PD. PD has been responsible for 30-62%, diarrhea associated deaths of young children in low- and middle- income countries. And in Bangladesh, PD accounted for more than 25% of all diarrhea related deaths among children aged 1-4 years and 40% of them were found malnourished.An international working group had developed and tested an algorithm through a multi country cohort for the treatment of PD nearly twenty years ago.However, this stepwise dietary algorithm increases the duration of hospital stay. To reduce the osmotic burden frequently children are given 3/4th strength diet. Though these diets are iso-osmolar, they provide suboptimal energy to the children. Several studies demonstrated the beneficial effect of green banana (GB) (whole green banana fruit, Musa paradisiacal sapientum) in the resolution of PD.The anti-diarrheal action of GB is postulated to be mediated by its high content of amylase-resistant starch (ARS), which is not digested in the small intestine of humans. On reaching the colon, it is fermented by resident bacteria into the short-chain fatty acids (SCFA) butyrate, propionate, and acetate. In the colon, SCFA stimulate salt and water absorption as well as provide energy and induce a trophic effect on the colonic as well as small-bowel mucosa. As 3/4th strength rice suiji is not providing sufficient calorie we are proposing to give full-strength rice suji as one intervention, and to ascertain the efficacy of GB in children suffering from undernutrition and/or co-morbidities we are proposing to give GB mix full strength rice suiji as another intervention.

Study design: This will be an open-labeled randomized controlled clinical trial with three treatment arms (3/4th strength rice suji, full strength rice suji with modification and GB mixed full strength rice suji). Investigators will prospectively screen, children > 6 to 36 months of age admitted to the Dhaka hospital of icddr,b, with PD or developed PD during their treatment period and failed to respond with milk suji and enroll them for the study. Thereafter permuted block randomization technique will be followed to select treatment arms for each child.

Study Area: The study will be conducted at the Dhaka hospital of the International Centre for Diarrheal Disease Research, Bangladesh (icddr,b), Dhaka, Bangladesh.This hospital provides care and treatment to over 140,000 patients annually of all ages and either sex, among them the number of under-five children were 83285. For critically ill patients there is an intensive care unit (ICU) facility present within the hospital, equipped with necessary life support measures including mechanical ventilators, syringe pump for vasopressor support.

Clinical management:

Usually children having PD will be admitted to the longer stay unit of the Dhaka hospital. An initial routine investigation will be done by the treating unit to identify the etiology of diarrhea whether infectious or noninfectious by doing stool RE and RS; TC, DC, Hb%. If stool RE suggestive of invasive diarrhea, appropriate antibiotic will be provided according to hospital protocol. During this period, milk suji, a low lactose diet, will be given as a routine diet. If child's PD resolved with milk suji, the child will be discharged with common health related advices. On day 4 (3 days after milk suji), if PD doesn't resolve, the child will be enrolled in the study and randomization will be done. The child will get either of the three diets- green banana mixed full strength rise suji, full strength rice suji, or 3/4th strength rice suji. With any of these diets, a child will be followed for 7 days. If there is deterioration of diarrhea (either increased frequency or watery consistency) for 3 days or condition remains static up to 7 days the child will be declared as treatment failure. Because this study duration will be for 7 days, after these one week of management, the child will not remain in the study and will receive standard management of the Dhaka hospital of icddr,b.

Sample size:

With 80 % power and 5% type I error and considering three treatment arms, Investigators need 40 children in each arm. If 45 children is enrolled in each arm,it will be able to accommodate up to 11 % attrition

So, the total sample size = 45*3= 135

ELIGIBILITY:
Inclusion Criteria:

* Children aged > 6 to 36 months, having diarrhea for 14 days or more (up to 29 days) either at admission or developed at some point during their treatment period in hospital
* Children able to take oral feeds at the time of randomization

Exclusion Criteria:

* Children whose parents/care givers do not provide consent
* Growth of Shigella, Salmonella or Cholera in rectal swab culture
* Children having WLZ/WHZ < -5 SD or +++ edema
* The children presented with septic shock, convulsion or any other illness that needs ICU support during the admission
* Birth defect like complex congenital heart diseases, cleft lip and cleft palate, Down syndrome and cerebral palsy and others that may itself cause digestive problem or failing to thrive
* Children diagnosed as having apparent or known tuberculosis or HIV or chronic (> 30 days)/organic diarrhea (where the cause is known e.g. crohn's disease, ulcerative colitis, celiac disease etc.)

Ages: 6 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 135 (Estimated)
Dates: Start 2017-12-07 (Actual); Primary Completion 2021-10-30 (Estimated); Study Completion 2021-10-30 (Estimated)

PRIMARY OUTCOMES:
By day 5, percentage of children recovered from diarrhea by the study diets | 5 days
  Recovery from diarrhea is desired in PD.so, study outcome will be measured by calculating the percentage of children recovered from diarrhea by the study diets by day 5.

SECONDARY OUTCOMES:
By day 7, percentage of children recovered from diarrhea by the study diets | 7 days
  Recovery from diarrhea is desired in PD. So, one of the secondary outcome is to find the percentage of children recovered from diarrhea by the study diets by day 7.
Frequency of stool in different days in different study diet groups | 7 days
  One of the study outcome is to record frequency of bowel movement whether reduced or increased.
Consistency of stool in different days in different study diet groups | 7 days
  One of the study outcome is to record stool consistency whether soft or formed.
Number of hospital acquired infection (HAI) in different study diet groups | 7 days
  At hospital, children are at risk of getting HAI, the number of HAI with different diet will be recorded.
Rate of relapse within 14 days follow up | 14 days
  If a child's PD resolved with study diet, the child will be discharged with the study diet. After discharge a child will be followed for 14 day with 2 follow up visit with the aim to identify the relapse rate.

CONTACTS AND LOCATIONS:
Overall Officials: Monira Sarmin, MBBS, Principal Investigator — Medical officer, ICU
Locations (1):
- Dhaka Hospital, icddr,b, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sarmin M, Hossain MI, Islam SB, Alam NH, Sarker SA, Islam MM, Chisti MJ, Islam SMR, Mahfuz M, Ahmed T. Efficacy of a Green Banana-Mixed Diet in the Management of Persistent Diarrhea: Protocol for an Open-Labeled, Randomized Controlled Trial. JMIR Res Protoc. 2020 Mar 6;9(3):e15759. doi: 10.2196/15759. PMID 32224490